CLINICAL TRIAL: NCT00876213
Title: Amylin and GLP-1: Influence on Gastric Emptying, Appetite and Food Intake in Humans.
Brief Title: Amylin and Glucagon-Like Peptide-1 (GLP-1): Influence on Gastric Emptying, Appetite and Food Intake in Humans
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: University of Copenhagen, University of Copenhagen
Other Study IDs: KA-20060095
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes
Keywords: Amylin; GLP-1; gastric emptying; appetite and food intake
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this proposal is to dissect the mechanisms controlling gastric emptying, appetite and food intake in humans, and to obtain new knowledge to fight obesity on a pharmacological basis.

DETAILED DESCRIPTION:
The objective of the present study is to elucidate the mechanisms behind the effects of glucagon-like peptide-1 (GLP-1) on gastric emptying, appetite and food intake. The first GLP-1 based anti-diabetic therapy was approved by the FDA in 2005 and is now on the market in the United States. The strong glucose-dependent insulinotropic property of GLP-1 is a highly attractive feature in the pursue of optimal glycaemic control in type 2 diabetes. Moreover, the potential of GLP-1 to reduce gastric emptying, appetite and food intake makes it an attractive tool in the fight against obesity, a pandemic condition that often leads to type 2 diabetes, and several companies are developing weight lowering drugs based on GLP-1. Interestingly, another peptide, amylin, exerts very similar effects on gastric emptying, appetite and food intake in humans. Amylin is found in insulin-rich granules in pancreatic beta-cells and is co-secreted with insulin upon insulinotropic stimuli. Currently, it is not known whether the inhibiting effects of GLP-1 on gastric emptying, appetite and food intake are directly mediated by GLP-1, or if the effects are secondary to the robust insulin responses, and thereby amylin responses, elicited by GLP-1. The objective of the present study is therefore to further elucidate the mechanisms of these effects in order to strengthen the development of anti-diabetic drugs with potential weight lowering capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes

  * Informed oral and written consent
  * Caucasians over the age of 18 years with type 1 diabetes (diagnosed according to the criteria of WHO) receiving long acting insulin
  * C-peptide negative glucagon test
  * Normal blood haemoglobin concentration
* Healthy control subjects

  * Informed oral and written consent
  * Caucasians over the age of 18 years
  * Normal 75 g- oral glucose tolerance test (OGTT) according to the criteria of WHO
  * Negative islet cell autoantibodies (ICA) and GAD-65 autoantibodies
  * No first-degree relatives with diabetes
  * Normal blood haemoglobin concentration

Exclusion Criteria:

* Patients with type 1 diabetes

  * Residual beta-cell function (evaluated with glucagon test)
  * Impaired hepatic function (aspartate aminotransferase (ASAT) and/or alanine aminotransferase (ALAT) > 2 times upper normal limit)
  * Diabetic nephropathy (serum-creatinine > 130 µM and/or albuminuria)
  * Diabetic neuropathy
  * Proliferative diabetic retinopathy
  * Pregnancy, breastfeeding or intention of becoming pregnant or judged to be using inadequate contraceptive measures
* Healthy control subjects

  * Impaired hepatic function (ASAT or ALAT > 2 times upper normal limit)
  * Impaired renal function (serum-creatinine > 130 μM and/or albuminuria)
  * First-degree relatives with diabetes
  * Pregnancy, breastfeeding or intention of becoming pregnant or judged to be using inadequate contraceptive measures

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with type 1 diabetes and matched healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-03; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meena Asmar, MD,Ph.Dstud., Principal Investigator — Panum Institut; Jens Juul Holst, Professor,MD, Study Director — Panum Institut
Locations (1):
- Hvidovre Hospital, Hvidovre, Hvidovre, Denmark